CLINICAL TRIAL: NCT00738790
Title: The Randomised Study of Preoperative Radiotherapy and Local Excision for Radiosensitive Rectal Cancer
Brief Title: Preoperative Radiotherapy and Local Excision in Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Colorectal Cancer Study Group (Network)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Poznan University of Medical Sciences (Other); Medical University of Lublin (Other)
Responsible Party: Prof. Marek P. Nowacki, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology in Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGBRJG0108; KBN0655/P05/2005/28
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; preoperative radiotherapy and local excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Preoperative radiotherapy with five fractions of 5 Gy during one week and boost 4 Gy after 1 week interval, total dose 29 Gy; after 6 weeks full-thickness local excision
  Interventions: Radiation: Short course of radiotherapy
- 2 (Active Comparator): Radiochemotherapy with 28 fractions of 1,8 Gy plus boost 5,4 Gy in 3 fractions
  + simultaneous bolus 5-Fluorouracil and leucovorin; after 6 weeks full-thickness local excision
  Interventions: Radiation: Radiochemotherapy

INTERVENTIONS:
Radiation: Short course of radiotherapy — 5 x 5 Gy plus boost 4 Gy
  Other Names: short radiation
  Arms: 1
Radiation: Radiochemotherapy — 28 x 1,8Gy plus boost 3 x 1,8 Gy with three 2-days cycles of chemotherapy during weeks 1, 3 and 5 of irradiation (the each cycle consisted of leukovorin 20 mg/m2 per day and 10-20 minutes later of 5-fluorouracil 400 mg/m2 per day, both administrated as rapid intravenous infusion)
  Other Names: chemoradiation
  Arms: 2

SUMMARY:
According to the current opinion, local excision in rectal cancer should be limited to selected T1N0 tumours. The investigators addressed the question whether preoperative radio(chemo)therapy can expand the use of this procedure for more advanced cancers. The rationale of preoperative radiotherapy is eradication of mesorectal subclinical disease. Besides, there is a correlation between radiosensitivity of rectal cancers and low cancer aggressiveness. For this reason, conversion to abdominal surgery is needed in patients with radioresistant tumour. The investigators aim to compare the short-course radiotherapy schedule with the chemoradiation in order to determine an optimal scheme. The study hypothesis is that the chemoradiation assures 25% more patients who do not require conversion to an open surgery. In addition, the aim is to asses safety and efficiency of preoperative radiotherapy and local excision for radiosensitive rectal cancer.

DETAILED DESCRIPTION:
Local excision must involve all tissue invaded on pretreatment examination. For this reason, 4-5 tatoos of mucosa at the tumour border should be performed before the onset of treatment. Next, the long-course radiochemotherapy or short-course radiotherapy is randomly allocated. After 6 weeks interval, the full thickness local excision should be carried out with 1 cm margin. Patients with good pathological response (complete response or downstaging to ypT1 disease)are followed up. Conversion to open surgery is offered to patients with poor pathological response (ypT2-3 or positive margin). Close follow-up is carried out in order to detect an early local recurrence either in a bowel wall or in mesorectal lymph nodes. Rescue surgery is offered in patients with local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven good or moderately differentiated adenocarcinoma of rectum
* Extraperitoneal tumour (< 3-4 cm; unfavourable cT1 or cT2-3; N0)
* No evidence of distant metastases on chest X-ray and abdominal CT or sonography
* Signed by patient written informed consent

Exclusion Criteria:

* Poorly differentiated pathology (G3)
* Patients unfit for chemotherapy
* No agreement for randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2003-11; Primary Completion 2010-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with downstaging after radiotherapy to pathological complete response or ypT1 disease with negative margins. | Surrogate endpoint available immediatly after surgery.

SECONDARY OUTCOMES:
The rate of local control, overall survival and disease-free survival and toxicity. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bujko, Prof., Principal Investigator — Roentgena 5, 02-781 Warsaw, Poland
Locations (1):
- M. Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland

REFERENCES:
- [Background] Bujko K, Sopylo R, Kepka L. Local excision after radio(chemo)therapy for rectal cancer: is it safe? Clin Oncol (R Coll Radiol). 2007 Nov;19(9):693-700. doi: 10.1016/j.clon.2007.07.014. Epub 2007 Sep 4. PMID 17766096
- [Background] Bujko K, Richter P, Kolodziejczyk M, Nowacki MP, Kulig J, Popiela T, Gach T, Oledzki J, Sopylo R, Meissner W, Wierzbicki R, Polkowski W, Kowalska T, Stryczynska G, Paprota K; Polish Colorectal Study Group. Preoperative radiotherapy and local excision of rectal cancer with immediate radical re-operation for poor responders. Radiother Oncol. 2009 Aug;92(2):195-201. doi: 10.1016/j.radonc.2009.02.013. Epub 2009 Mar 16. PMID 19297050